CLINICAL TRIAL: NCT06034496
Title: Cranial Electrotherapy Stimulation (CES) Influences on Acute Stress Responses
Brief Title: Cranial Electrotherapy Stimulation and Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00003572
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anxiety State
Keywords: Cranial Electrotherapy Stimulation; Acute Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Coded devices with master key kept outside of research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active CES (Active Comparator): Active Cranial Electrotherapy Stimulation (CES)
  Interventions: Device: Active CES
- Sham CES (Sham Comparator): Sham Cranial Electrotherapy Stimulation (CES)
  Interventions: Device: Sham CES

INTERVENTIONS:
Device: Active CES — Active CES group will receive a minimum of 250µA and up to 500µA depending on thresholding, once daily for 20 days (over the course of 4~6 weeks), 20 minutes per day.
  Other Names: Alpha-Stim
  Arms: Active CES
Device: Sham CES — Sham CES group will be identical to Active CES group with the exception of the device not administering any electrical current
  Other Names: Alpha-Stim
  Arms: Sham CES

SUMMARY:
The goal of this study is to quantify the effects of 20 sessions of Cranial Electrotherapy Stimulation (CES) on measures of acute stress responses in Soldiers. The main question it aims to answer is how 20 sessions of CES will affect Soldiers' biochemical (salivary alpha amylase and cortisol), physiological (e.g., heart rate, heart rate variability, respiration rate), emotional (state anxiety), and behavioral (i.e., cognitive task performance) responses.

* On Day 1, participants will complete a baseline measure assessing their biochemical, physiological, emotional, and behavioral responses to a stressful lethal force decision making task.
* In the next four to six weeks, participants will complete 20 CES sessions.
* Within five days of completing the 20 CES sessions, participants will complete a follow-up measure assessing their biochemical, physiological, emotional, and behavioral responses to the same stressful lethal force decision making task they completed on Day 1.

Researchers will compare the Active CES group to the Sham CES group to see how 20 sessions of Active CES will affect the participants responses to their biochemical, physiological, emotional and behavioral responses relative to the Sham CES group.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age (17-40 if emancipated minor)
* Can sit and stand freely.
* Have not used or experienced CES administration in the past.
* Agree to have their data stored in a repository (database) for future use.

Exclusion Criteria:

* Use of prescription medications, other than oral contraceptives
* Women only:

  1. Pregnant or plan to become pregnant during the study
  2. Nursing
* History of:

  1. A neurological or psychological disorder (such as depression, anxiety disorders, migraines, cluster headaches, seizures, Post-traumatic stress disorder (PTSD) or panic attacks).
  2. Cardiac disease (including arrhythmia or fast or skipped heart beats).
  3. Implanted medical devices, such as pacemakers.
  4. Hypertension.
  5. Insomnia
  6. Head injury (including neurosurgery, concussion, TBI, skull fracture, hematoma)
  7. Illness that caused brain injury
  8. Any other brain-related condition (such as traumatic brain injury)
  9. Metal in the head (outside of mouth, such as shrapnel, surgical clips, or fragments from welding or metalwork)
  10. Implanted medical device (e.g., pacemaker, insulin pump)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kana Okano, Ph.D., Principal Investigator — Tufts University
Locations (1):
- Tufts University, Medford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participants consent to having their deidentified data placed in a repository/shared upon protocol closure, however it is not mandated by the protocol or institution.

REFERENCES:
- [Derived] Okano K, Lee MM, Hart-Pomerantz H, Smith M, Sandone MK, Harvey T, Brunye TT. Effects of repeated cranial electrotherapy stimulation on physiological and behavioral responses to acute stress: a double-blind randomized clinical trial. Front Hum Neurosci. 2025 Aug 13;19:1641801. doi: 10.3389/fnhum.2025.1641801. eCollection 2025. PMID 40881935

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 participants consented to participate in the study. However, 18 participants (soldiers) were unable to start the study due to scheduling conflicts. Therefore, only 58 are included in the Participant Flow.
Period: Overall Study
Arm/Group | Active CES | Sham CES
Started | 28 | 30
Completed | 21 | 25
Not Completed | 7 | 5
Not completed — Did not meet minimum stimulation threshold | 2 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CES | Sham CES | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.95 (2.94) | 23.36 (5.82) | 22.26 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 25 | 46
Education [Mean (Standard Deviation); unit: years] | 13.95 (1.43) | 14.6 (3.04) | 14.3 (2.44)
STAI-T [Mean (Standard Deviation); unit: units on a scale] — State Trait Anxiety Inventory - Trait version
  units on a scale | 33.71 (10.75) | 29.52 (7.28) | 31.43 (9.17)
Military [Count of Participants; unit: Participants] | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Heart Rate During Stressful Lethal Force Decision Making Task
Description: heart rate will be measured in beats per minute.
Time Frame: Baseline and follow-up session after 20 CES to be completed within 4-6weeks
Population: Due to technical issues, we were unable to collect data from 9 participants.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 18 | 19
bpm
  Baseline | 98.5 (16.1) | 111 (19.5)
  Follow-up | 100.0 (13.5) | 114 (20.1)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .012, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .33, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .85, ANOVA — Session (baseline, follow-up) x CES

2. Primary Outcome: Change From Baseline in Respiration Rate During Stressful Lethal Force Decision Making Task
Description: respiration rate will be measured in breaths per minute.
Time Frame: Baseline and follow-up session after 20 CES to be completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: breath per minute
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 18 | 19
breath per minute
  Baseline | 16.2 (3.52) | 17.7 (3.53)
  Follow-up | 17.3 (3.05) | 16.8 (3.22)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .6, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .9, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .05, ANOVA — CES x Session interaction

3. Primary Outcome: Change From Baseline in Heart Rate Variability During Stressful Lethal Force Decision Making Task
Description: Heart rate variability will be measured in RMSSD.
Time Frame: Baseline and follow-up session after 20 CES to be completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 18 | 19
bpm
  Baseline | 13.0 (5.17) | 11.2 (4.53)
  Follow-up | 12.0 (4.76) | 10.5 (4.74)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .26, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .17, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .73, ANOVA — CES x Session main effect

4. Primary Outcome: Change Over Time in Cortisol During Stressful Lethal Force Decision Making Task
Description: Cortisol (µg/dL) will be measured through saliva samples. Saliva samples will be taken at five time points, approximately 20 minute increments during the baseline and follow-up sessions.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 21 | 25
µg/dL
  Baseline Pre | .293 (.137) | .415 (.183)
  Baseline 0min post | .54 (.36) | .399 (.105)
  Baseline 20min post | .57 (.396) | .655 (.476)
  Baseline 40min post | .371 (.194) | .456 (.252)
  Baseline 60min post | .29 (.156) | .369 (.197)
  Follow-up Pre | .335 (.149) | .345 (.123)
  Follow-up 0min post | .644 (.433) | .556 (.296)
  Follow-up 20min post | .444 (.206) | .534 (.292)
  Follow-up 40min post | .407 (.268) | .417 (.163)
  Follow-up 60min post | .335 (.198) | .379 (.171)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .18, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — Time main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .53, ANOVA — CES main effect
Statistical Analysis 4: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .07, ANOVA — CES x Time interaction
Statistical Analysis 5: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .46, ANOVA — CES x Session
Statistical Analysis 6: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .01, ANOVA — Time x Session interaction
Statistical Analysis 7: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .29, ANOVA — CES x Time x Session interaction

5. Primary Outcome: Change Over Time in Alpha Amylase During Stressful Lethal Force Decision Making Task
Description: Alpha amylase (IU) will be measured through saliva samples. Saliva samples will be taken at five time points, approximately 20 minute increments during the baseline and follow-up sessions.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 21 | 24
IU
  Baseline Pre | 118 (90.6) | 79.1 (69.2)
  Baseline 0min post | 144 (91.3) | 131 (121)
  Baseline 20min post | 88.6 (50.6) | 84 (61)
  Baseline 40min post | 110 (87.6) | 78.1 (58.2)
  Baseline 60min post | 105 (66.2) | 79.8 (61.2)
  Follow-up Pre | 68.4 (51.0) | 61.7 (48.6)
  Follow-up 0min post | 99.8 (39.3) | 129 (101)
  Follow-up 20min post | 110 (71.8) | 90.8 (72.6)
  Follow-up 40min post | 91.2 (49.5) | 92.6 (78.6)
  Follow-up 60min post | 128 (84.9) | 97.5 (91.7)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .10, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — Time main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .81, ANOVA — Session main effect
Statistical Analysis 4: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .40, ANOVA — CES x Time interaction
Statistical Analysis 5: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .35, ANOVA — CES x Session interaction
Statistical Analysis 6: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — Time x Session interaction
Statistical Analysis 7: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .40, ANOVA — CES x Time x Session interaction

6. Primary Outcome: Change Over Time in State Trait Anxiety Inventory (STAI) Scores at Each Session From Baseline to Follow-up
Description: STAI assesses both state and trait anxiety separately with each scale ranging from 20 to 80, with higher scores correlating with greater anxiety. STAI-S is the State Trait Anxiety Inventory - State version, and STAI-T is the State Trait Anxiety Inventory - Trait version.
Time Frame: At baseline, at each of the 20 CES sessions completed within 4-6weeks, and at follow-up to be completed within 5 days of last CES
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 21 | 25
score on a scale
  STAT-T at baseline Pre CES intervention | 33.71 (10.75) | 29.52 (7.28)
  STAT-T at follow-up Post CES intervention | 33.33 (12.72) | 32.64 (7.16)
  STAI-S Baseline Session Pre-Stress task | 33.4 (7.94) | 31.0 (6.62)
  STAI-S Baseline Session 0min Post Stress task | 39.5 (10.7) | 41.6 (12.2)
  STAI-S Baseline Session 20min Post Stress task | 35.6 (11.5) | 34.1 (9.53)
  STAI-S Baseline Session 40min Post Stress task | 32.4 (9.79) | 30.6 (8.54)
  STAI-S Baseline Session 60min Post Stress task | 30.9 (9.56) | 29.1 (6.66)
  STAI-S Follow-up Session Pre Stress task | 33.8 (15.0) | 27.6 (8.55)
  STAI-S Follow-up Session 0min Post Stress task | 34.6 (12.0) | 33.0 (10.8)
  STAI-S Follow-up Session 20min Post Stress task | 30.4 (11.6) | 29.3 (8.55)
  STAI-S Follow-up Session 40min Post Stress task | 29.0 (9.95) | 26.6 (7.94)
  STAI-S Follow-up Session 60min Post Stress task | 29.1 (9.75) | 26.1 (8.13)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .23, ANOVA — STAI-T CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .45, ANOVA — STAI-T Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .38, ANOVA — STAI-T CES x Session interaction
Statistical Analysis 4: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .40, ANOVA — STAI-S CES main effect
Statistical Analysis 5: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — STAI-S Time main effect
Statistical Analysis 6: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — STAI-S Session main effect
Statistical Analysis 7: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .20, ANOVA — STAI-S CES x Time interaction
Statistical Analysis 8: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .39, ANOVA — STAI-S CES x Session interaction
Statistical Analysis 9: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — STAI-S Session x Time interaction
Statistical Analysis 10: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .38, ANOVA — STAI-S CES x Time x Session interaction

7. Primary Outcome: Change From Baseline in Recognition Memory
Description: Recognition memory of previously learned targets while ignoring visually similar distractor objects will be measured and evaluated with percent accuracy.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: percent accuracy
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 17 | 21
percent accuracy
  Baseline | 77.1 (11) | 80 (12.2)
  Follow-up | 78.2 (15.9) | 76.7 (14.3)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .85, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .69, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .4, ANOVA — CES x Session interaction

8. Primary Outcome: Change From Baseline in Spatial Orientation
Description: Spatial orientation task will involve pointing towards a series of distant (out of visible range) landmarks in the virtual environment and estimating distance to those landmarks. Spatial orientation will be calculated using mean absolute angular error. Larger numbers correlate with higher error.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: absolute angle error in degrees
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 19 | 21
absolute angle error in degrees
  Baseline | 20.7 (8.12) | 18.8 (10.4)
  Follow-up | 21.2 (12.7) | 16.3 (10.1)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .13, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .26, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .44, ANOVA — CES x Session interaction

9. Primary Outcome: Change From Baseline in Decision Making Accuracy
Description: Participants will make lethal force decision making by shooting at threatening targets and allowing non-threatening targets to pass. Decision making accuracy will be calculated using d prime. Higher d prime correlates with better accuracy.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Measure: Mean (Standard Deviation); unit: d prime
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 17 | 20
d prime
  Baseline | 3.64 (.681) | 3.89 (1.08)
  Follow-up | 4.48 (.943) | 4.75 (1.29)
Statistical Analysis 1: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .36, ANOVA — CES main effect
Statistical Analysis 2: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .00, ANOVA — Session main effect
Statistical Analysis 3: Comparison: Active CES vs Sham CES; Test type: Superiority; p = .96, ANOVA — CES x Session interaction

10. Primary Outcome: Change From Baseline in Decision Making Reaction Time
Description: Participants will make lethal force decision making by shooting at threatening targets and allowing non-threatening targets to pass. Decision making reaction time to shoot at threatening targets will be measured in milliseconds.
Time Frame: Baseline and follow-up session after 20 CES completed within 4-6weeks
Population: Collected data were invalid and could not be analyzed due to a coding error. The coding error incorrectly summed and aggregated the distances of all avatars on the screen, rather than isolating the distance of the specific avatar that was shot. As a result, we were unable to reverse engineer the output to derive a value that accurately reflected Reaction Times.
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | Active CES | Sham CES
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 2/28 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 0.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active CES (N=28) | Sham CES (N=30)
Dizziness (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This research is funded by the U.S. Special Operations Command (SOCOM). Disclosure of research findings is subject to government operational security (OPSEC) and Public Affairs Office (PAO) review processes, in accordance with DoD Directives 5205.02E and 5230.29. As such, the Principal Investigator's ability to publicly disseminate or discuss trial results following study completion is restricted until appropriate clearances are obtained.

DOCUMENTS (3):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT06034496/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT06034496/SAP_004.pdf
  • Informed Consent Form (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT06034496/ICF_001.pdf